CLINICAL TRIAL: NCT06362915
Title: Analgesic Effect of Illiohypogastic & Ilioinguinal Nerve Block in TAVR - TF (Prospective Randomized Study)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, maha sadek El Derh, Assistant professor of Anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASUR66/2024
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: Anesthesia, Local
MeSH Terms: interventions — Lidocaine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: * Group (A): will receive blind local infiltration in femoral region on the operation side by an experienced anesthesiologist using 20 ml lidocaine 1% (9).
  * Group (B): will receive ultrasound-guided ilioinguinal/iliohypogastric nerve block using 20 ml Bupivicane 0.25% by an experienced anesthesiologist.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A:Lidocaine group (Active Comparator): will receive blind local infiltration in femoral region on the operation side by an experienced anesthesiologist using 20 ml lidocaine 1%
  Interventions: Drug: Lidocaine
- Group B:Bupivacaine group (Active Comparator): will receive ultrasound-guided ilioinguinal/iliohypogastric nerve block using 20 ml Bupivicane 0.25% by an experienced anesthesiologist
  Interventions: Drug: Bupivacain

INTERVENTIONS:
Drug: Lidocaine — * Group (A) lidocaine : will receive blind local infiltration in femoral region on the operation side by an experienced anesthesiologist using 20 ml lidocaine 1%.
  Arms: Group A:Lidocaine group
Drug: Bupivacain — • Group (B),bupivacaine: will receive ultrasound-guided ilioinguinal/iliohypogastric nerve block using 20 ml Bupivacaine 0.25% by an experienced anesthesiologist
  Arms: Group B:Bupivacaine group

SUMMARY:
The purpose of the study is to compare the effect of illiohypogastric and ilioinguinal nerve block with the local infiltration with lidocaine in patients undergoing TAVI

DETAILED DESCRIPTION:
This prospective, randomized, double blinded study will take place at cardiothoracic academy, Ain Shams University hospitals, Cairo, Egypt. In this study, participants, care providers and outcomes assessors will be ignorant of the treatment allocation. The study will start after obtaining the ethical approval & will continue for a 1 year. All patients will sign written informed consent before inclusion.

Patients fulfilling criteria for TAVI regarding age & pathology of aortic valve will be included in the study.

Exclusion criteria:

Refusal of the patients, Patients with neurological disease (Disturbed conscious level or psychiatric illness) severe respiratory disease need mechanical ventilation or need respiratory support, coagulation abnormalities, infection at site of injection.

After confirming the diagnosis & preoperative sizing of the valve by CT heart and then confirmation that no need for TEE guidance of the procedure, we will include 60 patients and then will be divided into two groups according to the technique of local anesthesia for the site of puncture.

Sample size calculation was done using G power program; setting power at 80% and α error at 5%, a sample size 52 patients undergoing transcatheter aortic valve implantation "TAVI" (26 patients receiving iliohypogastric with ilioinguinal nerve block and 26 patients receiving local infiltration with lidocaine) will be added to detect a statistically significant difference between the two groups as regard analgesic consumption, assuming a large effect size difference (dz=0.8)regarding Hasak et al.,2019. Patients will be randomly allocated into two equal groups each one made of 30 patients, the allocation ratio is 1:1 and the method of randomization will be computer generated randomized numbers, and it will be hidden in sealed opaque envelopes to conceal the allocation. The study will start after acquisition of ethical approval and expected to continue for a year.

* Group (A): will receive blind local infiltration in femoral region on the operation side by an experienced anesthesiologist using 20 ml lidocaine 1%.
* Group (B): will receive ultrasound-guided ilioinguinal/iliohypogastric nerve block using 20 ml Bupivicane 0.25% by an experienced anesthesiologist. (9).

In both group all patients undergo preoperative assessment: Full history, examination & investigations.

ECG, ECHO, CT heart and CT coronary angiography, LL venous & arterial duplex, CBC, Kidney and liver functions, Coagulation profile & carotid duplex.

Inside the catheterization room, for both groups after standard monitors and invasive hemodynamic monitors were applied (US guided arterial in left radial, CVC inserted in left IJV & sheath in right IJV for pacemaker).

Then Dexmedetomidine started in both groups by 0.1 up to 0.5 mic/kg/hour without loading with continuous monitoring for the HR and BP .

Then the patients divided into two groups: group for local infiltration and group for ilioinguinal illiohypogastric nerve block.

During injection of local anesthesia in both group any hemodynamic changes (blood pressure and heart rate should be closely monitored and recorded during data collection.

TAVI procedure will be proceeded. All patients were sent to ICU for postoperative care. HR, MAP, Conscious level of the patient assessed every 5 minutes. Need for increments narcotics or Propofol recorded and collected at end of procedure.

A Study made in 2019 on the effect of illiohypogastric ilioinguinal nerve block in TAVI patient found that Ultrasound-guided II-IH nerve block produce better intraoperative analgesia and less analgesic consumption than local infiltration anesthesia in patients undergoing TAVI .

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling criteria for TAVI regarding age & pathology of aortic valve will be included in the study.

Exclusion Criteria:

Refusal of the patients, Patients with neurological disease (Disturbed conscious level or psychiatric illness) severe respiratory disease need mechanical ventilation or need respiratory support, coagulation abnormalities, infection at site of injection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-07-15 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Extra Demand of sedation | All through procedure
  Need for increments of narcotics or propofol will be recorded and collected at the end of the procedure.

SECONDARY OUTCOMES:
Patient and surgeon satisfaction | all through the procedure
  Patient satisfaction in form not complaining or asking for more analgesic or deepen anesthesia.
  Surgical satisfaction in form of quiet noncomplaining patient, hemodynamic stability

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - maha sadek El Derh, Cairo, Heliopolis
  - Ain Shams University, Cairo

IPD SHARING:
Plan to Share IPD: No